CLINICAL TRIAL: NCT05086484
Title: Omics Sequencing of Specimen Derived From Patients With Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZhujiangHfck
Record Dates: First submitted 2021-10-01; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Endometriosis
Keywords: Endometriosis; microbiota; metabolomic
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis group: Women diagnosed with endometriosis.
- Control group: Women diagnosed without endometriosis.

SUMMARY:
Endometriosis is a type of chronic inflammatory gynecological disease, mainly took place in peritoneal cavity. In order to investigate the possible correlation between microbes and endometriosis, the investigators planed to perform 16S rDNA amplicon sequencing, metagenomic sequencing and metabolomic sequencing of paired samples derived from feces, cervical mucus, blood and peritoneal fluid.

ELIGIBILITY:
Inclusion Criteria:

1. The subject who is female.
2. The subject who is infertility or sub-fertile.
3. The subject whose age was between 18-52 years old.
4. The subject who is suspected to have endometrioma.
5. The subject whose menstrual cycle length is between 28-35 days.
6. The subject without the history of abdominal or pelvic surgery.
7. The subject who has dysmenorrhea.
8. The subject who has dispareunia.
9. The subject who was informed the risks and benefits of the experiment and provided written informed consent, and gave their approval.
10. The subject who has chronic pelvic pain and the pain get worse during periods.
11. The subject who has no sexual activity within a week.
12. The subject who has no history of acute or chronic pelvic inflammatory disease.
13. The subject who has confirmed EM with biopsy.
14. The subject without hormonotherapy within 6 months.
15. The subject without medical history of antibiotics within 6 months.

Exclusion Criteria:

1. The subject who has hernia.
2. The subject who is pregnant.
3. The subject who has malignant tumor.
4. The subject who has Gene Therapy history.
5. The subject who has abdominal or pelvic surgery history.
6. The subject who has peritonitis.
7. The subject who is below 18 years old or over 52 years old.
8. The subject who can not endure laparoscopy.
9. The subject who has cardiovascular disease.
10. The subject who has systemic or regional acute inflammation.
11. The subject who has chronic liver or kidney disease.
12. The subject whoes body mass index ≤ 18.5 or ≥ 28 (kg m-2).
13. The subject who has coagulation defects or hematologic diseases.
14. The subject who has tuberculosis or chronic obstructive pulmonary disease.
15. The subject whoes alcohol consumption ≥ 60 g d-1, or smokers (≥20 cigarettes d-1).
16. The subject who has hypertension, diabetes, hyperthyroidism and ect.
17. The subject whoes medical history of transfusion, stem cell or bone marrow transplantation.
18. The subject who has contraindication of tracheal intubation anesthesia.
19. The subject who received hormonotherapy within 6 months.
20. The subject who has immunodeficient, allergic or autoimmune diseases.
21. The subject who used antibiotics within 6 months.
22. The subject who is drug abuse.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women at reproductive age.
Study Population: Study population are those who are admitted to Zhujiang Hospital of Southern Medical University in Guangzhou, China, due to gynecological diseases. At least two gynecologists independently screened and assessed the condition of the participants strictly according to the inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
16s amplicon sequencing | 2019/01/01-2023/12/31
  Compare the microbiota composition differences of specimens derived from control group and Endometriosis group.
metatranscriptomic sequencing | 2019/01/01-2023/12/31
  Compare the RNA concentration differences of specimens derived from control group and Endometriosis group.
metabolomic sequencing | 2019/01/01-2023/12/31
  Compare the metabolites concentration differences of specimens derived from control group and Endometriosis group.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China